CLINICAL TRIAL: NCT04627844
Title: Ideal Time to Enteral Feeding Following Percutaneous Endoscopic Gastrostomy Tube Placement
Brief Title: Time to Feeding After PEG Tube Placement.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Andrew Lawson, Assistant Professor, Trauma/Critical Care, General Surgery, Augusta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1656460-1
Record Dates: First submitted 2020-09-25; First posted 2020-11-13 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Feeding Tube Complication

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive feeding beginning at two time points.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Delayed Feeds (Placebo Comparator): Patients will receive tube feeds beginning at 6 hours after PEG tube placement. This is our institutions current practice
  Intervention Type: Dietary
  Interventions: Dietary Supplement: Delayed Feeding
- Immediate Feeds (Experimental): Patients will receive tube feeds beginning immediately after PEG tube placement.
  Intervention Type: Dietary
  Interventions: Dietary Supplement: Immediate Feeding

INTERVENTIONS:
Dietary Supplement: Immediate Feeding — Standard tube feeds begun at an earlier time point
  Arms: Immediate Feeds
Dietary Supplement: Delayed Feeding — Standard tube feeds begun at delayed time point
  Arms: Delayed Feeds

SUMMARY:
Trauma patients who require Percutaneous Endoscopic Gastrostomy (PEG) tube placement for feeding and who consent to be in the study will be randomized to receive feeding at either 6 hours after PEG placement as is routinely done or at 0 hours after PEG placement.

DETAILED DESCRIPTION:
Critically ill patients share a common hypermetabolic response to injury, deterioration in lean body mass, and a high rate of septic complications. Route of nutrition administration influences the response to injury. A well-fed intestine absorbs nutrients while maintaining an effective barrier against pathogens, added by adequate peristalsis, mucin production, and immunoglobulin A secretion. In critical care patients, enteral nutritional therapy (EN) feeding has been shown to restores normal gut architecture and microflora, improve the immune system response, and aid the mucosa in withstanding insult to the system. Studies have shown that those on EN feeding have reduced morbidity and mortality rates as well as fewer infections and have less line-associated sepsis when compared to parenteral nutritional therapy (PN) feeding.

There are multiple EN feeding methods. Percutaneous endoscopic gastrostomy (PEG) was first introduced in 1980, and due to PEG being low cost, minimally invasive, and having no need for Bernal anesthetic in most cases, it is considered a better choice for the introduction of feeding than other methods. PEG tubes are usually entered for periods of tube feeding lasting more than 30 days, as well as when a nasogastric tube cannot but used for nutritional support. However, compared to naso-enteric tubes, PEG tubes are associated with fewer complications, greater patient comfort, better aesthetic appearance, and improved patient quality of life. For this reason, PEG is currently the method of choice for medium- and long- term enteral feeding. Previous studies have found complication rates within 30 days of PEG tube placement to be 10-15%.

Traditionally, post-PEG insertion, feeding was delayed until the next day for fear of peritoneal leakage risk after feeding. However, multiple studies have shown that feeding after PEG can be started early, within hours without a significant increase in the procedure-related morbidity or mortality and thereby reducing the healthier costs. There is currently no standard of practice for the timing of enteral feeding following PEG placement. Each group has different practice guidelines, and no national consensus has been established.

Studies have indicated that the initiation of tube feeding three to four hours after an uncomplicated PEG was safe, well-tolerated, and helped to reduce the hospital stay. A systematic analysis of five studies found that there were no significant differences between enteral feeds beginning at 3 hours versus feeds beginning at later times.

The investigator's current institution does not have a standard of practice for time to begin feeding after PEG tube placement; that decision is currently provider dependent. A survey of providers at the investigator's institutions indicated that the most common time to begin feeds is 6 hours, however, providers at the institution use varied times to beginning feeds between 0 and 24 hours after placement. The current literature supports a reduction in complications at feeds beginning under four hours. In fact, all studies investigating shorter time to feeds have found no associated increase in complications. No study to date has investigated immediately beginning tube feeds. There is no national consensus regarding feeding time after placement. Given the shown benefits of early enteral nutrition on reducing mortality and complications across a variety of conditions, the investigators believe early feeding has the strong potential to improve patient morbidity and mortality following PEG tube placement. This study aims to investigate whether beginning feeds immediately is a safe and effective management option for patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who require PEG tube placement for feeding by the Trauma/Acute Care Surgery at our institution who are able to provide consent or whose legally authorized representative is able to provide consent for the patient.

Exclusion Criteria:

* Patients not receiving PEG placement
* Patients receiving PEG tube placement by a member of a different hospital service
* Patients under the age of 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Severe complication | Typically up to 4 weeks
  Number of patients with a complication requiring return to operating room

SECONDARY OUTCOMES:
Minor complication | Through study completion, an expected average of one year
  Number of patients with a complication requiring cessation of feeds

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bechtold ML, Matteson ML, Choudhary A, Puli SR, Jiang PP, Roy PK. Early versus delayed feeding after placement of a percutaneous endoscopic gastrostomy: a meta-analysis. Am J Gastroenterol. 2008 Nov;103(11):2919-24. doi: 10.1111/j.1572-0241.2008.02108.x. Epub 2008 Aug 21. PMID 18721239
- [Background] Choudhry U, Barde CJ, Markert R, Gopalswamy N. Percutaneous endoscopic gastrostomy: a randomized prospective comparison of early and delayed feeding. Gastrointest Endosc. 1996 Aug;44(2):164-7. doi: 10.1016/s0016-5107(96)70134-7. PMID 8858322
- [Background] Cristian D, Poalelungi A, Anghel A, Burcos T, Grigore R, Bertesteanu S, Richiteanu G, Grama F; -. Prophylactic Percutaneous Endoscopic Gastrostomy (PEG) - The Importance of Nutritonal Support in Patients with Head and Neck Cancers (HNCs) or Neurogenic Dysphagia (ND). Chirurgia (Bucur). 2015 Mar-Apr;110(2):129-36. PMID 26011834
- [Background] Kudsk KA, Croce MA, Fabian TC, Minard G, Tolley EA, Poret HA, Kuhl MR, Brown RO. Enteral versus parenteral feeding. Effects on septic morbidity after blunt and penetrating abdominal trauma. Ann Surg. 1992 May;215(5):503-11; discussion 511-3. doi: 10.1097/00000658-199205000-00013. PMID 1616387
- [Background] McCarter TL, Condon SC, Aguilar RC, Gibson DJ, Chen YK. Randomized prospective trial of early versus delayed feeding after percutaneous endoscopic gastrostomy placement. Am J Gastroenterol. 1998 Mar;93(3):419-21. doi: 10.1111/j.1572-0241.1998.00419.x. PMID 9517650
- [Background] Rahnemai-Azar AA, Rahnemaiazar AA, Naghshizadian R, Kurtz A, Farkas DT. Percutaneous endoscopic gastrostomy: indications, technique, complications and management. World J Gastroenterol. 2014 Jun 28;20(24):7739-51. doi: 10.3748/wjg.v20.i24.7739. PMID 24976711
- [Background] Szary NM, Arif M, Matteson ML, Choudhary A, Puli SR, Bechtold ML. Enteral feeding within three hours after percutaneous endoscopic gastrostomy placement: a meta-analysis. J Clin Gastroenterol. 2011 Apr;45(4):e34-8. doi: 10.1097/MCG.0b013e3181eeb732. PMID 20733512